CLINICAL TRIAL: NCT06119074
Title: Assessing the Impacts of a Novel Unconditional Gifted Savings Program
Brief Title: A Novel Unconditional Gifted Savings Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project did not receive expected funding.
Sponsor: University of Pennsylvania (Other)
Collaborators: Universal Gifted Savings (Unknown)
Responsible Party: Principal Investigator, Stacia West, Associate Professor & Co-Founding Director of the Center for Guaranteed Income Research, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 854513
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Poverty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gifted Savings (Experimental): Participants in the treatment group will receive an unconditional Gifted Savings account with $2,000 of assets ($100 USD available upon enrollment; $500 USD available for emergency use each year for two years).
  Interventions: Other: Gifted Savings
- No Gifted Savings (No Intervention): Participants in the control group will not receive a Gifted Savings account.

INTERVENTIONS:
Other: Gifted Savings — Gifted Savings assets will be in the form of cash, Bitcoin, and/or stock. Participants will receive identical asset portfolios. The asset mix will be determined by Gifted Savings. Participants will not have any control over the assets they receive, nor the proportion of each in their account. After registration on the Gifted Savings website, participants can immediately withdraw $100 USD if they choose. Then, for each of the first two years, participants may withdraw up to $500 USD for an emergency (self-attested) if the value of the account is 50% or more of its value 30 days prior and the account has sufficient funds to fulfill the request. Two years post-enrollment, participants may withdraw the entire value of their GS account or continue holding the assets in their GS account (in perpetuity or until the GS non-profit ceases to exist). GS funds are unconditional; there are no restrictions or limitations on how the money can be spent.
  Arms: Gifted Savings

SUMMARY:
The goal of this randomized control trial is to test the impacts of an unconditional Gifted Savings account of $2,000 of assets ($100 United States Dollars available upon enrollment; $500 United States Dollars available for emergency use each year for two years) on adults with household incomes of three times the Federal Poverty Level or less in Yellow Springs, Ohio.

DETAILED DESCRIPTION:
Many lower to middle income families are unable to weather an unforeseen financial emergency. Even in the best economic conditions, the personal saving rate in the US is profoundly low: just under 10% of disposable income. The consequences are as follows:

* Some low to middle income families, and particularly families of color and those headed by single women, turn to alternative financial services (pawn shops, credit cards not paid in full, high-interest loans, and payday lenders) to cover the financial shock. Others turn to family and friends.
* Over time, and with constrained financial resources, some households are unable to pay back these alternative financial services resulting in substantial debt. In the event these households turn to family and friends on a recurrent basis, relationships and a person's sense of dignity, worth, and control over one's future are fractured.
* These financial conditions cause stress, anxiety, and other mental health issues that lock a person in the here and now--rationally occupied with the dire economic conditions of the present and unable to plan for the future This has a resultant impact on cognitive capacity, hope for the future, future savings and goals horizons, and mental well-being.

This randomized control trial is being conducted to evaluate a program created by Gifted Savings (GS), an experimental non-profit start-up. GS is not a bank or an insured financial institution. GS will issue accounts seeded with $2,000 of assets in the form of cash, Bitcoin, and/or stock the experimental study group (n=250). The control group (n=500) will not receive a GS account but will be invited to complete study surveys every six months for 36 months.

For participants who receive a GS account, the original value of the account is not guaranteed, as assets may increase or decrease in value over time depending on market conditions. After two years, participants may withdraw the entire value of their GS account or choose to continue holding the assets in the GS account. Assets may be held forever or until the GS non-profit ceases to exist. GS funds are unconditional, which means there are no restrictions or limitations on how the money can be spent. Withdrawn funds will be available by check or direct deposit.

Over three years, researchers will measure the impacts of receiving a Gifted Savings account on:

* Psychological distress
* Employment and income
* Financial well-being
* Agency and hope for the future
* Material hardship
* Savings behavior and horizons
* Ability to manage financial shocks
* Subjective financial knowledge
* Cryptocurrency knowledge, attitudes, and behaviors

All participants will complete:

* A baseline survey
* Follow-up surveys at 6-, 12-, 18-, 24-, 30-, and 36-months after enrollment

Participants who receive a Gifted Savings account will:

* Register on the Gifted Savings website to claim their account
* Hold their Gifted Savings account assets for at least two years

Some participants who receive a Gifted Savings account will also participate in an in-depth interview.

Researchers will compare participants who receive a Gifted Savings account to participants who do not receive a Gifted Savings account to test the effects of receiving a Gifted Savings account on the above research questions.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Yellow Springs, Ohio
* At least 18 years of age
* Annual household income of three times the Federal Poverty Level or less

Exclusion Criteria:

* Not a resident of Yellow Springs, Ohio
* Under 18 years of age
* Annual household income of more than three times the Federal Poverty Level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Financial-well being (Consumer Financial Protection Bureau Financial Well-Being Scale) | 6 months
  Each item is scored 0 to 4 and summed to a total. The sum total is then converted to a total response value on the CFPB Financial Well-Being Scale score from 0-100.
Financial shock | 6 months
  Five items to assess participants' ability to cover a $400 emergency expense, frequency of $400 emergency expenses over past 6 months, length of time savings could sustain household, likelihood of finding $2,000 for emergency expense, and estimated savings needed for future emergency expenses.
Savings | 6 months
  Eight items to assess bank account ownership status (yes/no), savings and investing behaviors, past month's amount saved, total amount saved, confidence about meeting future financial obligations, and savings horizons.
Stress and coping (Perceived Stress Scale - 4) | 6 months
  Each item is scored from "never" to "all of the time" on a 5-point scale. Scores of 4 items are then summed, yielding a minimum score of 0 and a highest score of 16. Higher scores are correlated to more stress.
Mental health (Kessler 10) | 6 months
  Each item is scored from one "none of the time" to five "all of the time." Scores of the 10 items are then summed, yielding a minimum score of 10 and a maximum score of 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress.
Hope (Adult Hope Scale) | 6 months
  Four items measure pathways thinking, four items measure agency thinking, and four items are fillers. The four pathways thinking items and the four agency thinking items are scored from one "definitely false" to eight "definitely true," then summed for a total score. Higher scores indicate higher levels of hope.
Financial confidence | 6 months
  Two items to assess confidence in household's ability to meet longer term goals and comfort with current financial situation.
Liabilities | 6 months
  Eleven items to assess: past 6 month use of shadow banking services (e.g., check cashing, payday loans, auto title loans), late fees charged, spending compared to income, credit score (very bad to very good/I don't have a credit score/I don't know), types of debt, and debt payments.
Housing hardship | 6 months
  Three items from the U.S. Census Bureau's Survey of Income and Program Participation to assess rent/mortgage payments, recent eviction, and utility payments/disconnections.

SECONDARY OUTCOMES:
Relational finances | 6 months
  Three items to assess past month provision of financial help to family or friends, amount loaned, and reason for loan. Three items to assess past month receipt of financial help from family or friends, amount borrowed, and reason for borrowing.
Employment status | 6 months
  Three items to assess current employment status, educational status, and occupation type.
Subjective financial knowledge | 6 months
  Answer to single-item question: "On a scale from 1 to 7, where 1 means very low and 7 means very high, how would you assess your overall financial knowledge?" (1 is very low; 7 is very high).
Cryptocurrency knowledge, attitudes, and behaviors | 6 months
  Six items to assess participants' experiences with cryptocurrency.
Mastery (Pearlin Mastery Scale) | 6 months
  This seven-item scale includes five negatively worded items and two positively worded items. Each item is scored from one "Strongly Disagree" to four "Strongly Agree." The negatively worded items are reverse coded. Scores are summed, resulting in a score range of 7 to 28, with higher scores indicating greater levels of mastery.
Food insecurity | 6 months
  Answer to single item question "In the past 6 months, I worried whether our food would run out before I got money to buy more" (often; sometimes; rarely; never).

OTHER OUTCOMES:
Website usability | 12 months
  Answer to the single-item Net Promotor Score question: "How likely are you to recommend Gifted Savings to a friend or relative?" (0 not likely to 10 very likely), and the two-item "UX-LITE" scale, scored from strongly disagree (1) to strongly agree (5), where higher summed scores means better usability.

CONTACTS AND LOCATIONS:
Overall Officials: Stacia West, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No